CLINICAL TRIAL: NCT00799214
Title: Back to BASICS: Boric Acid, Alternate Solution for Intravaginal Colonization, Comparing Intravaginal Metronidazole to Boric Acid in Women Symptomatic for Bacterial Vaginosis
Brief Title: BASIC (Boric Acid, Alternate Solution for Intravaginal Colonization) Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H07-02330
Record Dates: First submitted 2008-11-10; First posted 2008-11-27 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Bacterial Vaginosis
Keywords: bacterial vaginosis; intravaginal; boric acid; metronidazole; placebo controlled; double-blind; randomized; multicenter; non-inferiority
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — boric acid; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): 1 gram emollient cream to be inserted intravaginally qhs (once before bed) for 10 days or less if intolerable side effects occur.
  Interventions: Drug: Placebo
- 2 (Experimental): Boric acid = 600 mg boric acid compounded in emollient cream (1 gram total) to be inserted intravaginally qhs (once before bed) for 10 days or less if intolerable side effects occur.
  Interventions: Drug: Boric acid
- 3 (Active Comparator): Metronidazole = 10 % intravaginal cream (Sanofi-Aventis Canada Inc Product DIN 01926861) (for a total of 37.5 mg metronidazole) inserted intravaginally qhs (once before bed) for 10 days or less if intolerable side effects occur.
  Interventions: Drug: Metronidazole

INTERVENTIONS:
Drug: Placebo — 1 gram emollient cream to be inserted intravaginally qhs (once before bed) for 10 days or less if intolerable side effects occur.
  Arms: 1
Drug: Boric acid — Boric acid = 600 mg boric acid compounded in emollient cream (1 gram total) to be inserted intravaginally qhs (once before bed) for 10 days or less if intolerable side effects occur.
  Arms: 2
Drug: Metronidazole — Metronidazole = 10 % intravaginal cream (Sanofi-Aventis Canada Inc Product DIN 01926861) (for a total of 37.5 mg metronidazole) to be inserted intravaginally qhs (once before bed) for 10 days or less if intolerable side effects occur.
  Arms: 3

SUMMARY:
Bacterial vaginosis (BV), the world's most common vaginal infection, continues to cost patients time, energy, comfort and money. BV is associated with increased incidence of sexually transmitted infections (including HIV), spontaneous abortion, pre-term labour, post-surgical infections, and endometritis. Current treatment for those women symptomatic for BV includes both oral and intravaginal antibiotics, such as metronidazole, which have success rates of 70-80 % at 1 month after treatment. These treatments also have high recurrence rates (49-66 % at one year after treatment) and side effects (10-20 % of women) that include secondary vaginal infection with candida. Intravaginal boric acid has been used for >100 years for the treatment of vaginal infections and is quite commonly prescribed today as a treatment for BV. It is cheap, easily accessible, easy to use, and is an effective treatment of other vaginal infections, such as candida. To date, there are no clinical trials studying the effectiveness of boric acid in the treatment of BV.

The objective of this study was to determine whether intravaginal BA is comparable to standard treatment, metronidazole, for the cure of BV in symptomatic women.

Our research question is: Among women 16-50 years old symptomatic with BV is intravaginal treatment with BA non-inferior to metronidazole to achieve a Nugent score <7 (cure) by day 17.

Hypothesis: H0: BA proportion of women cured < metronidazole proportion of women cured - 10%.

DETAILED DESCRIPTION:
A minimum of 240 volunteer women will be recruited through participating family practice offices throughout British Columbia. Women with symptoms of BV, who also have a positive whiff test/pH test or subsequent positive vaginal swab for BV, will be asked to participate. Women will be included if they have both a positive test result for BV (whiff test/vaginal swab) and if they have any symptoms of BV present. The following criteria must be met for enrolment in the study: 1) ages 16-50 and pre-menopausal; 2) capable of giving written informed consent; 3) fluent comprehension of spoken and written English; 4) negative pregnancy test on enrolment day; 5) agree to follow study protocol; 6) documented BV infection by positive vaginal swab (minimum Nugent score of 7/10) +/- positive whiff test/pH >4.5; 7) agree to no intercourse for the 10 days of treatment (or to use non-lubricated condoms if unavoidable); 8) agree not to douche or use any intravaginal products during treatment (including tampons, medications, devices); 9) abstain from alcohol during the 10 days of treatment (from 24 hours before through 72 hours after taking study medication); 10) agree to no new medications or antibiotics during treatment; 11) no current sexually transmitted infection as determined by history, physical exam and negative swabs for chlamydia, gonorrhea, candidiasis, trichomonas; 12) patient is reliable for follow up.

The following women would be excluded from study participation: 1) less than 16 or post-menopausal; 2) menstruating at diagnosis; 3) symptoms so severe as to make allocation to placebo unacceptable to the patient; 4) currently pregnant or at high risk for pregnancy; 5) current sexually transmitted infection (HIV, hepatitis, chlamydia, gonorrhea, trichomonas, HPV or HSV); 6) current yeast infection as determined by history, physical and swabs; 7) history of PID; 8) allergy to latex or metronidazole; 9) presently breast feeding; 10) any open wound, excoriation, vaginal irritation and including bartholin's cyst/abscess as determined by physical exam; 11) presence of another vulvar, vaginal or medical condition, including cervical neoplasia/treatment, that might confound treatment response; 12) using lithium, anti-coagulants or disulfiram drugs; 13) any antifungal or antibiotic use 14 days prior to enrolment 14) PAP smear done within one week of enrolment, 15) positive Whiff test, but negative vaginal swab result.

During the initial visit, the physician will take a history and do a speculum and manual pelvic exam for the woman. At the time of the pelvic exam the physician will ensure intact mucous membranes and anatomy, take swabs for chlamydia and gonorrhea, bacterial vaginosis, candidiasis, and trichomonas, and perform a whiff test using a provided, standardized 10% KOH potassium hydroxide solution. Vaginal discharge will also have pH testing done. If the whiff test is positive and the vaginal discharge pH is >4.5, the woman will then take a urine pregnancy test, will be informed about the study, and will be given a handout explaining the study and the 3 possible treatment arms.

If the woman is interested in participating she will be given a "Study Intake Survey" to fill out, a consent form to sign, and an assigned number.

Within a few days, the physician would confirm participation, eligibility and exclusion criteria and collect the signed consent form. The patient will then be given a blinded, controlled and randomized treatment pack containing 10 capsules compounded and organized by a pharmacist. The patient will be given a package containing: 1) capsule applicators; 2) pads; 3) non-lubricated condoms; 4) a diary to record their daily use of the treatment, any problems or side effects, any symptom changes, or any problems with maintaining the study agreements; 5) information sheet outlining follow up instructions and emergency contact numbers to reach the study members. If the woman does not want to join the study the physician will prescribe a standard treatment of their choosing and would follow up as usual. If the whiff test is negative but the vaginal swab is found to be positive for bacterial vaginosis as per the Nugent score (score minimum of 7/10), the woman will be called back in to the office. If her symptoms are found to be persistant at this juncture, then she will be offered to enroll in the study or may elect to start a treatment of her physician's choosing. If the woman prefers to take some time to decide about the study, she will be given the information package, the survey form, and consent form to take home, as well as a prescription for the treatment of bacterial vaginosis. She can then return the next day with the forms filled out should she decide she would like to enroll in the study and be assigned a treatment arm. If she chooses not to enroll, she can fill the above-mentioned prescription and start the treatment for BV provided by her physician.

The women who satisfy the inclusion and exclusion criteria will be blindly and randomly assigned to one of 3 treatments (minimum of 80 women per treatment arm): 1) placebo (emollient cream); 2) boric acid (600 mg boric acid in emollient cream); 3) metronidazole 10 % intravaginal cream (Sanofi-Aventis Canada Inc Product DIN 01926861) (for a total of 37.5 mg metronidazole) ). The treatments will be taken at night prior to sleep using the provided applicators for 10 days. The patient will be instructed to use a provided pads during the day and night for any discharge or fluid. The patient will record daily in a diary (provided) about compliance, side effects and problems, and changes in symptoms over the 10 days. The patient will be welcome to call the provided emergency numbers of the study members for any questions or problems related to the treatment. On day 5 of the treatment, the patient will receive a call or email from a study member to ask follow up questions about compliance, side effects, BV symptoms, and satisfaction of treatment.

On both follow up visits: days 17-19 (one week after the treatment end) and 40-42 (one month after the treatment end), the participant will return to the clinic that enrolled her for reassessment, pregnancy test, and follow up examination including pelvic exam and repeat swabs. It will be noted whether her BV symptoms are still present, and if she had any side effects or problems during treatment. The participant returns her daily treatment diary on day 17 visit as well.

ELIGIBILITY:
Inclusion Criteria:

Women will be included whether their complaint is symptoms of BV and have a positive whiff test/vaginal swab or if they have a positive whiff test/vaginal swab and are then asked if they have any symptoms of BV present. The following criteria must be met for enrolment in the study:

1. ages 16-50 and premenopausal;
2. capable of giving written informed consent;
3. English speaking;
4. negative pregnancy test on enrolment day;
5. agree to follow study protocol;
6. documented BV infection by positive vaginal swab +/- positive whiff test/pH > 4.5;
7. agree to no intercourse for the 10 days of treatment (or to use non-lubricated condoms if unavoidable);
8. agree not to douche or use any intravaginal products during treatment (including tampons, medications, devices);
9. abstain from alcohol during the 10 days of treatment (from 24 hours before through 72 hours after taking study medication);
10. agree to no new medications or antibiotics during treatment;
11. no current sexually transmitted infection as determined by history, physical exam and negative swabs for chlamydia, gonorrhea, candidiasis, trichomonas;
12. patient is reliable for follow up.

Exclusion Criteria:

The following women would be excluded from study participation:

1. less than 16 or post-menopausal;
2. negative vaginal swab regardless of whiff test/pH > 4.5;
3. menstruating at diagnosis;
4. symptoms so severe as to make allocation to placebo unacceptable to the patient;
5. currently pregnant or at high risk for pregnancy;
6. current sexually transmitted infection (HIV, hepatitis, chlamydia, gonorrhea, trichomonas, HPV or HSV);
7. current yeast infection as determined by history, physical and swabs;
8. history of PID;
9. allergy to latex or metronidazole;
10. presently lactating;
11. any open wound, excoriation, vaginal irritation and including bartholin's cyst/abscess as determined by physical exam;
12. presence of another vulvar, vaginal or medical condition, including cervical neoplasia treatment, that might confound treatment response;
13. using lithium, anti-coagulants or disulfiram drugs;
14. any antifungal or antibiotic use 14 days prior to enrolment
15. PAP smear done within one week of enrollment.

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2014-04; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Non-inferiority, per protocol comparison of effectiveness of boric acid to metronidazole at day 17 as measured by Nugent score in 16-50 year olds with a z-based confidence interval for the difference of two proportions | day 17

SECONDARY OUTCOMES:
Non-inferiority, intent-to-treat comparison of effectiveness of boric acid to metronidazole at day 17 as measured by Nugent score in 16-50 year olds with a z-based confidence interval for the difference of two proportions | day 17
Non-inferiority, comparison of effectiveness of boric acid to metronidazole at day 40 as measured by Nugent score in 16-50 years old analyzed both per protocol and intent-to treat with a z-based confidence interval for the difference of two proportions | day 40
Safety consideration including intolerable adverse effects requiring patient discontinuation of the 10 day treatment | day 1-10

CONTACTS AND LOCATIONS:
Overall Officials: Konia Trouton, MD, Principal Investigator — University of British Columbia; Melinda Zeron Mullins, MD, Ph.D, Principal Investigator — University of British Columbia
Locations (1):
- Multicentered, family practice offices, Province-wide, British Columbia, Canada

REFERENCES:
- [Derived] Zeron Mullins M, Trouton KM. BASIC study: is intravaginal boric acid non-inferior to metronidazole in symptomatic bacterial vaginosis? Study protocol for a randomized controlled trial. Trials. 2015 Jul 26;16:315. doi: 10.1186/s13063-015-0852-5. PMID 26210791